CLINICAL TRIAL: NCT03657420
Title: A Phase Ib Investigation of the Safety and Efficacy of ABI-009 (Nab-rapamycin) in Combination With Pomalidomide and Dexamethasone for Relapsed and Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of ABI-009 (Nab-rapamycin) in Combination With Pomalidomide and Dexamethasone for Relapsed and Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn by sponsor
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-252
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABI-009 + Pomalidomide + Dexamethasone (Experimental): * Pomalidomide is given orally daily on days 1-21, 7 days off
  * ABI-009 is given intravenously on days 1, 8, and 15
  * Dexamethasone is given orally weekly on days 1, 8, 15, 22
  Interventions: Drug: ABI-009; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: ABI-009 — ABI-009 is an mTOR inhibitor. This pathway is believed to be overactive in multiple myeloma.
  Other Names: nab-rapamycin
Drug: Pomalidomide — Pomalidomide is an immunomodulatory agent and believed to work by affecting the growth signals that keep cancer cells alive.
  Other Names: Pomalyst
Drug: Dexamethasone — Dexamethasone is a steroid which is believed to kill cancer cells
  Other Names: Decadron

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for multiple myeloma.

The drugs that will be administered are:

* ABI-009 (nab-rapamycin)
* Pomalidomide
* Dexamethasone

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved ABI-009 as a treatment for any disease.

The FDA has approved pomalidomide and dexamethasone as treatment options for multiple myeloma.

The purpose of this study is to determine whether ABI-009 (study drug) will be safe and slow the progress of the disease when used in combination with pomalidomide and dexamethasone, depending on what type of cancer.

ABI-009 is an inhibitor of an overactive biological pathway in the cancer cells. Pomalidomide is an immunomodulatory agent and believed to work by affecting the growth signals that keep cancer cells alive. Dexamethasone is a steroid which is believed to kill cancer cells. The investigators hope that the combination of ABI-009 with pomalidomide and dexamethasone will help stop the growth of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated relapsed and refractory multiple myeloma. Relapsed and refractory is defined per International Myeloma Working Group Criteria (Rajkumar et al., 2011).
* Patients must have received at least two prior therapies with at least 2 cycles of lenalidomide and at least 2 cycles of a proteasome inhibitor (either in separate regimens or within the same regimen)
* Disease progression on or within 60 days of completion of last therapy.
* All laboratory assessments should be performed within 21 days of initiation of protocol therapy unless otherwise specified.
* Participant has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (see Appendix A).
* Age ≥ 18 years
* Measurable disease of multiple myeloma as defined by at least one of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL
  * ≥ 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum free light chain ≥ 100 mg/L (10 mg/dL) and abnormal serum free kappa to serum free kappa light chain ratio
* ANC ≥ 1000/μL. G-CSF is not permitted within 14 days of screening.
* Platelet count ≥ 75,000/µL. Platelet transfusions are not permitted within 7 days of screening.
* Hemoglobin ≥ 8 g/dL. Red blood cell transfusions are permitted to meet eligibility criteria.
* Calculated creatinine clearance of ≥ 30 mL/min according to Cockroft-Gault equation
* Patient has adequate hepatic function, as evidenced by the following:

  * Serum bilirubin values < 2 mg/dL, and serum alanine transaminase (ALT), and serum aspartate transaminase (AST) values < 3 × the institutional upper limit of normal (ULN).

Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval

* Must be able to take acetylsalicylic acid (ASA) daily as prophylactic anticoagulation. Patients intolerant to ASA may use low molecular weight heparin or equivalent. Warfarin will be allowed provided patient is fully anticoagulated, with an INR of 2-3.
* All study participants must be registered into the mandatory POMALYST REMS program and be willing and able to comply with the requirements of the POMALYST REMS program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the POMALYST REMS program.
* Able to swallow capsules whole (pomalidomide capsules cannot be crushed, dissolved or broken).

Exclusion Criteria:

* Prior therapy with mTOR inhibitor (e.g. everolimus, sirolimus). Note, prior pomalidomide therapy is permitted.
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the first dose or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier. Patients may have received dexamethasone within 2 weeks prior to entering study.
* Patients who are receiving any other investigational agents.
* Concomitant high dose corticosteroids except participants may be on chronic steroids (maximum dose 10 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, e.g. adrenal insufficiency, rheumatoid arthritis, etc.
* Pregnant or lactating females
* Prior history of malignancies, other than MM, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Ductal carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T1a or T1b)
* Patients undergoing active treatment for another malignancy with the exception of non-melanoma skin cancer or in situ cervical cancer.
* Patients with plasma cell leukemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) syndrome, or amyloidosis are excluded from this trial.
* HIV infection
* Active hepatitis B infection or active hepatitis C infection, per treating investigator. Patients who have prior hepatitis C infection but who have received an antiviral treatment and show no detectable viral RNA for 6 months are eligible
* Peripheral neuropathy ≥ grade 2 despite supportive therapy
* Hypersensitivity to thalidomide, lenalidomide, pomalidomide, bortezomib, or dexamethasone (such as Stevens-Johnson syndrome). Rash to immunomodulatory drug that can be medically managed is allowed
* Patients who had allogeneic stem cell transplant fewer than 12 months prior to initiation of study treatment and who have not discontinued immunosuppressive treatment for at least four weeks prior to initiation of study treatment and are currently dependent on such treatment.
* Patients with active graft v. host disease.
* History of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness that could preclude study participation, pose an undue medical hazard, or interfere with the interpretation of the study results, including, but not limited to, patients with congestive heart failure (New York Heart Association [NYHA] Class 3 or 4); unstable angina; cardiac arrhythmia; recent (within the preceding 6 months) myocardial infarction or stroke; hypertension requiring > 2 medications for adequate control; diabetes mellitus with > 2 episodes of ketoacidosis in the preceding 12 months; or chronic obstructive pulmonary disease (COPD) requiring > 2 hospitalizations in the preceding 12 months.
* Patient has any other medical, psychiatric, or social condition that would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results.
* History of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
* Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfanidine) within the 14 days prior to receiving the first dose of ABI-009.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose. | 1 Cycle (28-Days)
  The maximum Tolerated Dose (MTD) is the highest dose of ABI-009 (nab-rapamycin) when administered in combination with pomalidomide and dexamethasone that dose not cause unacceptable side effects. The maximum tolerated dose is determined in clinical trials by testing increasing doses on different groups of people until the highest dose with acceptable side effects is found. A standard 3+3 dose escalation design will be used to assess the MTD.

SECONDARY OUTCOMES:
Overall response rate. | 2 years
  The number of participants that achieve a partial response or better. This is assessed using International Myeloma Working Group criteria.
Progression free survival. | 2 years
  Progression free survival is defined as the time to disease progression or death from any cause, censored at date last known progression free for those who have not progressed or died. Progression is assessed using International Myeloma Working Group Criteria.
Treatment-emergent adverse events. | 2 years
  Adverse events will be assessed using CTCAE criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Yee, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No